CLINICAL TRIAL: NCT04036682
Title: A Phase 1/2, Open-Label, Multi-Center Trial to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of CLN-081 in Patients With Locally-Advanced or Metastatic Non-Small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutations Who Have Previously Received Platinum-Based Systemic Chemotherapy
Brief Title: A Phase 1/2 Trial of CLN-081 in Patients With Non-Small Cell Lung Cancer
Acronym: REZILIENT1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cullinan Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-081-001
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer; EGFR Exon 20 Mutation
Keywords: NSCLC; EGFR; Exon 20 insertions; CLN-081; TAS6417; zipalertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — zipalertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase 1 Dose Escalation (Accelerated Titration) (Experimental): CLN-081 BID in single patient dose escalation cohorts enrolling NSCLC patients with EGFR exon 20 insertion mutations that either have received or never received prior EGFR TKIs.
  Interventions: Drug: CLN-081
- Phase 1 Dose Escalation (Rolling Six) (Experimental): CLN-081 BID in Rolling Six dose escalation cohorts enrolling NSCLC patients with EGFR exon 20 insertion mutations.
  Interventions: Drug: CLN-081
- Phase 2a Dose Expansion(s) (Experimental): CLN-081 BID in expansion cohorts that may be opened at doses that meet pre-specified efficacy and safety criteria.
  Interventions: Drug: CLN-081
- Module A Food Affect (Experimental): Single-dose CLN-081 150 mg with and without high fat food intake.
  Interventions: Drug: CLN-081
- Module B (Experimental): CLN-081 BID in NSCLC patients with EGFR exon 20 insertion mutations that have received prior systemic therapy for locally advanced or metastatic disease.
  Interventions: Drug: CLN-081
- Module C (Experimental): CLN-081 BID to patients with EGFR exon 20 insertion mutant NSCLC after prior therapy with an agent approved for the treatment of ex20ins mutant NSCLC.
  Interventions: Drug: CLN-081

INTERVENTIONS:
Drug: CLN-081 — CLN-081 tablets
  Other Names: TAS6417; zipalertinib

SUMMARY:
CLN-081-001 is a Phase 1/2, open label, multi-center study of CLN-081 in patients with non-small cell lung cancer (NSCLC) harboring EGFR (epidermal growth factor receptor) exon 20 insertion mutations, to characterize the safety, determine the recommended Phase 2 dose (RP2D), and evaluate efficacy.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multicenter, first-in-human trial to evaluate the safety and tolerability, PK, PD, and efficacy of CLN-081 in patients with non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) exon 20 insertion mutations.

This trial is divided into multiple parts: Phase 1 Dose Escalation, Phase 2a Dose Expansion, Module A, Module B, and Module C.

The objectives of the dose escalation and dose expansion parts are to determine the safety, tolerability, recommended Phase 2 dose (RP2D), and preliminary anti-tumor activity of orally administered CLN-081 monotherapy.

The objective of Module A is to preliminarily assess the effect of food on the PK profile of CLN-081.

The objective of Module B is to further characterize the safety and efficacy of CLN-081 monotherapy in patients with EGFR exon 20 insertion mutation NSCLC who have received prior systemic anti-cancer treatment for locally advanced or metastatic disease.

The objective of Module C is to explore the safety, tolerability, and efficacy of CLN-081 monotherapy in patients with EGFR exon 20 insertion mutation NSCLC who have received prior treatment with an agent approved for EGFR exon 20 insertion mutant NSCLC

CLN-081 will be dosed twice daily (BID).

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (all patients).
2. Documented EGFR ex20ins mutation demonstrated by a validated test listed in Section 9.7 and performed in a Clinical Laboratory Improvement Amendments (CLIA)-certified or equivalent laboratory (all patients other than Module A Food Effect PK Assessment Module). Institutions that don't have access to these tests should contact the sponsor for assistance.
3. Prior treatment in the recurrent/metastatic disease setting including:

   1. A platinum-based chemotherapy regiment (or other chemotherapy regimen if platinum-based chemotherapy is contra-indicated)
   2. Any other approved standard therapy that is available to the patient, unless this therapy is contraindicated, intolerable to the patient, or is declined by the patient. In the case of a patient declining such therapy, documentation that the patient has been informed and declined should be documented in the medical record.
   3. No prior therapy is required for patients enrolled on Module A.
   4. Prior therapy with an agent approved by the local regulatory authorities for the treatment of EGFR ex20ins mutant NSCLC (Module C only).
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (except for patients enrolled on Module A).
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Ability to take pills by mouth.
8. Have the following laboratory values:

   1. Serum creatinine < 1.5 × upper limit of normal (ULN) or calculated creatinine clearance (CrCl) must be ≥ 50 mL/min/1.73 m2 (if calculated by Cockroft-Gault formula, the actual body weight must be used for CrCl unless body mass index [BMI] >30 kg/m2 then lean body weight must be used).
   2. Total bilirubin ≤ 1.5 × ULN unless prior history of Gilbert's syndrome.
   3. AST and ALT ≤ 2.5 × ULN, or ≤ 5 × ULN if due to liver involvement by tumor.
   4. Hemoglobin ≥ 9.0 g/dL in the absence of transfusion ≤ 14 days prior to the first dose of study drug on C1D1.
   5. Platelets ≥ 100 × 109 cells/L in the absence of transfusion <14 days prior to the first dose of study drug on Cycle 1 Day 1 (C1D1).
   6. Absolute neutrophil count ≥ 1.5 ×109 cells/L.
9. For Module A patients only: patients must have a negative coronavirus disease 2019 (COVID-19) polymerase chain reaction test prior to enrolment.
10. For Module B and Module C patients only: verification of suitable archived tumor tissue available at the participating center for biomarker analysis. A fresh biopsy is required if an archived sample is not available.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

R6, Phase 1 Expansion, Phase 2a, Module A and Module B Patients Only

1. Prior treatment with an EGFR ex20ins -targeting drug (eg, including, but not limited to poziotinib, mobocertinib, amivantamab, DZD9008, BDTX-189).

   Note: enrolment of patients treated previously with EGFR ex20ins-targeting drugs allowed selectively during accelerated titration dose escalation and Module C only.

   Module A Food Effect PK Assessment Module patients only
2. Conditions that compromise esophageal or gastrointestinal (GI) function, including esophageal, gastric, pancreatic, hepatobiliary, or small bowel carcinomas, or history of gastric resection.
3. Recurrent diarrhea, nausea, or vomiting.
4. Unable to refrain from or anticipates the use of:

   1. Any drug, including prescription and non-prescription medications, including drugs that change gastrointestinal motility (eg, loperamide) or gastric pH (eg, antacids, H2 antagonists, proton pump inhibitors), herbal remedies, or vitamin supplements within 14 days prior to the first dosing on Day 1 to follow-up.
   2. Any drugs known to be inhibitors or inducers of CYP3A enzymes and/or P-glycoprotein (P-gp), including St. John's Wort and grape fruit juice, within 28 days prior to the first dosing and throughout the PK assessment.
5. Any allergies to the composition of the high fat meal.
6. Patients who use tobacco products.

   All Patients
7. History of COVID-19-related pneumonitis requiring hospitalization.
8. History of COVID-19 infection within 4 weeks prior to enrolment, or clinically significant pulmonary symptoms related to prior COVID-19 pneumonitis.
9. Treatment with any of the following:

   1. An EGFR TKI ≤ 8 days or 5 × the terminal phase t1/2, whichever is longer, prior to the first dose of study drug on C1D1.
   2. Systemic anticancer treatment (excluding EGFR-TKIs as described above) within 14 days prior to the first dose of study drug on C1D1.
   3. Immunotherapy ≤ 28 days prior to the first dose of study drug on C1D1.
   4. Radiotherapy < 28 days and palliative radiation ≤ 14 days prior to the first dose of study drug on C1D1. If irradiated, lesions must have demonstrated clear-cut progression prior to being eligible for evaluation as target lesions.
   5. Major surgery (excluding placement of vascular access) ≤ 28 days of the first dose of study drug on C1D1.
10. Have any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia and skin pigmentation. Patients with chronic but stable Grade 2 toxicities may be allowed to enroll after agreement between the Investigator and Sponsor.
11. Have known or suspected leptomeningeal metastasis. Have known or suspected brain metastases or spinal cord compression, unless the condition has been asymptomatic, treated with surgery and/or radiation (if clinically indicated), and has been stable without requiring escalating corticosteroids or anti-convulsant medications for at least four weeks prior to the first dose of study drug on C1D1.
12. Prior therapy with CLN-081.
13. Known hypersensitivity to CLN-081 or any drugs similar in structure or class.
14. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, treatment-related pneumonitis, or any evidence of clinically active interstitial lung disease.
15. Cardiac conditions as follows: Patient has a history of congestive heart failure (CHF) Class III/IV according to the New York Heart Association (NYHA) Functional Classification or serious cardiac arrhythmias requiring treatment.
16. Resting QTcF > 470 msec.
17. Patient is unable to take drugs po due to disorders or diseases that may affect GI function, including but not limited to inflammatory bowel diseases (eg, Crohn's disease, ulcerative colitis) or malabsorption syndrome, or procedures that may affect gastrointestinal function, such as gastrectomy, enterectomy, or colectomy.
18. Have any condition or illness that, in the opinion of the Investigator, might compromise patient safety or interfere with the evaluation of the safety of the drug.
19. Pregnant or lactating females; females of child-bearing potential (FOCBP) must have a negative serum pregnancy test at within seven days prior to receiving study drug on C1D1. FOCBP and males with partners of child-bearing potential must agree to use adequate birth control (Section 16.3) throughout their participation and for six months following the last dose of study treatment.
20. History of another primary malignancy within 2 years prior to starting study drug on C1D1, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ.
21. Uncontrolled intercurrent illness including, but not limited to, uncompensated respiratory, cardiac, hepatic, or renal disease, active infection (including human immunodeficiency virus (HIV) and active clinical tuberculosis), or renal transplant; ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements.
22. For patients with a history of hepatitis B (HBV), negative PCR test is required. Patients with active hepatitis B (HBV) infection [as defined by a positive hepatitis B serum antigen (HBsAg) test and detectable HBV deoxyribonucleic acid (DNA)]. Patients ineligible due to detectable levels of HBV DNA at baseline may be rescreened for enrolment if their HBV DNA levels become undetectable after treatment with antiviral agents, and upon agreement between the Investigator and Sponsor.
23. For patients with a history of hepatitis C, active infection as defined by a reactive hepatitis C virus (HCV) antibody test and detectable HCV ribonucleic acid (RNA).
24. Active bleeding disorders.
25. The patient is, in the Investigator's opinion, unable or unwilling to comply with the trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
All Cohorts: The rate and severity of treatment emergent AEs. | 24 months
All Cohorts: The rate and severity of DLTs. | 24 months
Phase 2 Dose Expansion Cohorts: Overall response rate (ORR) | 24 months
Module A: Pharmacokinetic (PK) parameter | 24 months
  Maximum Plasma Concentration [Cmax]
Module A: Pharmacokinetic (PK) parameter | 24 months
  Area Under Curve [AUC]
Module B and C: Confirmed overall response rate (ORR) and duration of response (DOR) by independent review committee (IRC) | 24 months

SECONDARY OUTCOMES:
Phase 1 Dose Escalation and Expansion, Phase 2a Dose Expansion, and Module B and C Cohorts: ORR by Investigator assessment | 24 months
Phase 1 Dose Escalation and Dose Expansion, Phase 2a Dose Expansion, and Module B and C Cohorts: DOR (duration of response). | 24 months
Phase 1 Dose Escalation and Dose Expansion, Phase 2a Dose Expansion, and Module B and C Cohorts: DCR (disease control rate) | 24 months
Phase 1 Dose Escalation and Dose Expansion, Phase 2a Dose Expansion, and Module B and C Cohorts: PFS (progression free survival) | 24 months
Phase 1 Dose Escalation and Dose Expansion, Phase 2a Dose Expansion, and Module B and C Cohorts: OS (overall survival) | 24 months
All Cohorts: Assessment of maximum concentration (Cmax) | 24 months
All Cohorts: Assessment of area under curve (AUC) | 24 months
All Cohorts: Assessment of time to maximum concentration (tmax) | 24 months
All Cohorts: Assessment of terminal half-life (t1/2) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zosia Piotrowska, MD, Study Chair — Massachusetts General Hospital
Locations (64):
- United States (18):
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Pacific Shores Medical Group, Long Beach, California
  - AdventHealth, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Summit Medical Group PA, Florham Park, New Jersey
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - New York University Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Providence Cancer Center, Portland, Oregon
  - Providence Oncology & Hematology Care Clinic-Westside, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Cancer Specialists, Fairfax, Virginia
- Hong Kong University - Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliero Universitaria Careggi, Careggi
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I, Marche
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola
  - IRCCS-Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Modena, Modena
  - San Gerardo Hospital, Monza
  - Ospedale Santa Maria delle Croci, Ravenna
- Japan (7):
  - National Cancer Center Hospital East, Chiba
  - Niigata Cancer Center, Niigata
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo
- Netherlands (2):
  - The Netherlands Cancer Institute (NKI), Amsterdam
  - Leiden University Medical Center, Leiden
- Singapore (2):
  - Singapore Clinical Research Institute, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (9):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital (SNUBH), Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Asan Medical Center (AMC), Soeul
  - Korea University Guro Hospital, Soeul
  - Ajou University Hospital, Suwon
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon
- Spain (13):
  - University Hospital A Coruna, A Coruña
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Parc Tauli, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia l'Hospitalet, Barcelona
  - START Barcelona, Barcelona
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - University Hospital Quironsalud Madrid, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- Taiwan (5):
  - Chang Gung Medical Foundation Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piotrowska Z, Passaro A, Nguyen D, Ruiter G, Soo RA, Ho-Fun Lee V, Velcheti V, Tan DS, Lee SH, Kim SH, Wrangle J, Yang JC, Daga H, Juan Vidal OJ, Spira AI, Fernandez-Hinojal G, Kim SW, Umemura S, Provencio Pulla M, Keeton EK, Yang ZS, Li S, Xu ZC, Jones JA, Yu HA; REZILIENT1 Investigators. Zipalertinib in Patients With Epidermal Growth Factor Receptor Exon 20 Insertion-Positive Non-Small Cell Lung Cancer Previously Treated With Platinum-Based Chemotherapy With or Without Amivantamab. J Clin Oncol. 2025 Jul 20;43(21):2387-2397. doi: 10.1200/JCO-25-00763. Epub 2025 Jun 1. PMID 40450572
- [Derived] Piotrowska Z, Tan DS, Smit EF, Spira AI, Soo RA, Nguyen D, Lee VH, Yang JC, Velcheti V, Wrangle JM, Socinski MA, Koczywas M, Janik JE, Jones J, Yu HA. Safety, Tolerability, and Antitumor Activity of Zipalertinib Among Patients With Non-Small-Cell Lung Cancer Harboring Epidermal Growth Factor Receptor Exon 20 Insertions. J Clin Oncol. 2023 Sep 10;41(26):4218-4225. doi: 10.1200/JCO.23.00152. Epub 2023 Jun 29. PMID 37384848
- [Derived] Ye L, Chen X, Zhou F. EGFR-mutant NSCLC: emerging novel drugs. Curr Opin Oncol. 2021 Jan;33(1):87-94. doi: 10.1097/CCO.0000000000000701. PMID 33122578